CLINICAL TRIAL: NCT00808080
Title: A Clinical Trial of Cytotoxic T Cells Augmenting Autologous Hematopoietic Stem Cell Transplantation for Acute Myeloid Leukemia
Brief Title: A Clinical Trial of Cytotoxic T Cells Augmenting Autologous Hematopoietic Stem Cell (AHSC) Transplantation for Acute Myeloid Leukemia (AML)
Acronym: AMLCTL
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: lack of accrual
Sponsor: Thomas A. Lane, MD (Other)
Responsible Party: Sponsor-Investigator, Thomas A. Lane, MD, Professor of Pathology, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 070768
Record Dates: First submitted 2008-12-12; First posted 2008-12-15 (Estimated); Results first posted 2016-02-22 (Estimated); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: AML
Keywords: AML

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Biologic (Experimental): AML_CTL cells
  Interventions: Biological: AMLCTL

INTERVENTIONS:
Biological: AMLCTL — Ex-vivo expanded cytotoxic autologous AML-reactive T cells (CTL)

SUMMARY:
The aim of this protocol is to investigate a novel form of immune therapy for patients with acute myelogenous leukemia (AML) who are in remission (CR) but who are at high risk for relapse.

DETAILED DESCRIPTION:
Primary Aim: To conduct a Phase 1/2 clinical trial of autologous CTL-mediated immunotherapy in a homogeneous group of patients with AML who have recently received an autologous hematopoietic stem cell transplant. Specifically:

Phase 1: To determine the MTD of autologous AML-reactive cultured CTL in patients with AML who have recently received an AHSCT.

Phase 2: To determine 1 year progression-free survival of the study group vs institutional historical control group composed of a sequential series of recent patients who have received an AHSCT for AML.

ELIGIBILITY:
Inclusion Criteria (Initial Eligibility Screen):

* Diagnosis of AML, not M3
* At least 10% of circulating leukocytes are AML blast cells
* Age 18 through 75
* Sex male or female
* Patient is considered a potential candidate for AHSCT

Exclusion criteria (Initial Eligibility Screen):

* Participation in another immunotherapy trial within 30 days
* Presence of active malignancy other than AML
* History of autoimmune disease requiring systemic treatment
* ECOG performance status of 3 or 4
* Major organ system dysfunction
* Recent (30 days) or current use of steroids other than topical skin preparations
* History of allogeneic transplant
* Patients who, for any reason are not deemed candidates for AHSCT

Eligibility for autologous CTL Infusion:

Inclusion Criteria:

* Patient has CTL that are in sufficient number and are suitable for infusion
* Patient is stable, afebrile, engrafted, ECOG status 0-2, in CR and received AHSCT 45 - 60 days earlier.

Exclusion or delay criteria:

* Temperature > 38 C and/or known to be infected
* Absence of engraftment ANC > 500 and Plt > 20,000 unsupported
* Life expectancy less than 6 weeks
* Autoimmune disease requiring systemic treatment.
* ECOG performance status of 3 or 4
* Major organ system dysfunction

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Lane, MD, Principal Investigator — UCSD
Locations (1):
- UCSD, La Jolla, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Biologic: AML_CTL cells
  AMLCTL: Ex-vivo expanded cytotoxic autologous AML-reactive T cells (CTL)
  6 patients were enrolled, however none of the 6 patients became eligible to receive the AML CTL Infusion
Period: Overall Study
Arm/Group | Biologic
Started | 6
Completed | 0
Not Completed | 6
Not completed — Patients Became Ineligible for infusion | 6

BASELINE CHARACTERISTICS:
Arm/Group | Biologic
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6
Percent Circulating Blasts In Peripheral Blood [Mean (Full Range); unit: percentage of peripheral blood] | 52.7 [26 to 90]
Percent Blast Cells in Bone Marrow [Mean (Full Range); unit: percentage of bone marrow] | 67.4 [45 to 80]
WBC at Baseline [Mean (Full Range); unit: 1000 cells/mm^3] | 18.4 [4 to 66]
ANC at Baseline [Mean (Full Range); unit: 1000 cells/mm^3] | 2460.7 [480 to 7398]

OUTCOME MEASURES:

1. Primary Outcome: 6 Dose Cohorts for Safety Monitoring. Each Cohort is Assessed for DLT for One Month After Autologous Cultured CTL Infusion Prior to Enrolling the Next Cohort.
Time Frame: 2.5 years estimated
Population: Not Applicable as none of the enrolled patients became eligible for infusion
Arm/Group | Biologic
Number analyzed (Participants) | 0

2. Secondary Outcome: If Phase I Has Successfully Shown the Target Dose to be Below the MTD Continue Enrolling Until 38 Patients Have Received the Target Dose. Patients Will be Monitored for Safety and Efficacy.
Description: 6 patients were enrolled, however none of the 6 patients became eligible to receive the AML CTL Infusion. No CTL infusions were administered to any subject, consequently NO outcome measure results are available.
Time Frame: 2.5 years estimated
Population: None. 6 patients were enrolled, however none of the 6 patients became eligible to receive the AML CTL Infusion. No CTL infusions were administered to any subject, consequently NO outcome measure results are available.
Groups:
- Biologic: AML_CTL cells
  AMLCTL: Ex-vivo expanded cytotoxic autologous AML-reactive T cells (CTL)
  6 patients were enrolled, however none of the 6 patients became eligible to receive the AML CTL Infusion. NO CTL infusions were administered to any subject, therefore NO outcome measure results are available.
Arm/Group | Biologic
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: No adverse events or serious adverse events occurred related to study treatment as no patients have received their AML CTL infusion.
Arm/Group | Biologic
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Accrual trial was insufficient. No patient became eligible for CTL infusion. Cell culture information gleaned from a comparison of different culture methods will greatly facilitate future studies of autologous CTL-directed immunotherapy for AML.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No